CLINICAL TRIAL: NCT00007189
Title: Alzheimer's Disease Anti-Inflammatory Prevention Trial (ADAPT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: National Institute on Aging (NIA) (NIH); VA Puget Sound Health Care System (U.S. Federal Agency); University of Washington (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IA0026; U01AG015477 (NIH)
Record Dates: First submitted 2000-12-14; First posted 2000-12-14 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; Anti-inflammatory drugs
MeSH Terms: conditions — Alzheimer Disease | interventions — Naproxen; Celecoxib

INTERVENTIONS:
Drug: Naproxen Sodium (Aleve)
Drug: Celecoxib (Celebrex)

SUMMARY:
The purpose of this trial is to test the ability of the non-steroidal anti-inflammatory medications naproxen and celecoxib to delay or prevent the onset of AD and age-related cognitive decline.

DETAILED DESCRIPTION:
Considerable evidence suggests that inflammation may play a role in the neurodegenerative process of Alzheimer's disease (AD), and the use of non-steroidal anti-inflammatory drugs may be associated with reduced occurrence of AD. ADAPT is a randomized trial that will test the ability of the non-steroidal anti-inflammatory medications naproxen and celecoxib to delay or prevent the onset of AD and age-related cognitive decline. This long-term trial will run for 5 to 7 years.

The study is sponsored by the National Institute on Aging and is being conducted at the Roskamp Institute in Tampa, FL; the Veterans Affairs Puget Sound Health Care System with the University of Washington, in Seattle, WA; Boston University School of Medicine, in Boston, MA; the Johns Hopkins Medical Institutions, in Baltimore, MD; Sun Health Research Institute, in Phoenix, AZ; and the University of Rochester, in Rochester, NY. At each of these six sites, the goal is the enroll approximately 700 men and women, totalling 2,625 participants. Participants must be 70 years of age or older, have a parent, brother, or sister who has, or had, serious age-related memory loss, senility, dementia, or Alzheimer's disease.

Participants will be asked to take an anti-inflammatory medication or placebo (inactive pill) twice daily. Before enrolling in the trial, participants will be asked to go to a study site for two medical evaluations. Once enrolled, they will need to go to a study site for a medical evaluation every six months and to participate in a telephone interview twice a year for an average of up to seven years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older.
* Family history of parent, brother, or sister who has, or had, serious age-related memory loss, senility, dementia, or Alzheimer's disease.
* Study partner available to provide information on the cognitive status of the participant and to assist with monitoring of trial medications, if needed.
* Sufficient fluency in written and spoken English to participate in study visits and neuropsychological testing.
* Willingness to limit use of the following for the duration of the study: vitamin E (at doses greater than 400 IU per day), non-aspirin NSAIDs, histamine H2 receptor antagonists (Tagamet, for example), corticosteroids, anti-inflammatory or analgesic doses of aspirin (greater than 81 mg per day), Ginkgo biloba extracts
* Ability and intention to participate in regular study visits, in the opinion of the study physician.
* Provision of informed consent.

Exclusion Criteria:

* History of peptic ulcer disease with bleeding or obstruction.
* Clinically significant liver or kidney disease.
* History of hypersensitivity to aspirin, ibuprofen, celecoxib, naproxen, or other NSAIDs.
* Use of anti-coagulant medication.
* Cognitive impairment or dementia.
* Current alcohol abuse or dependence

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2625
Dates: Start 2001-01; Primary Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Breitner, MD, MPH, Principal Investigator — Professor and Head, Division of Geriatric Psychiatry, University of Washington School of Medicine; and Director, GRCC, VA Puget Sound Health Care System, Seattle
Locations (6):
- United States (6):
  - Sun Health Research Institute, Sun City, Arizona
  - Roskamp Institute Memory Clinic, 10770 N. 46th Street, Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Rochester, Rochester, New York
  - Veterans Affairs Puget Sound Health Care System, University of Washington, Seattle, Washington

REFERENCES:
- [Background] Anthony JC, Breitner JC, Zandi PP, Meyer MR, Jurasova I, Norton MC, Stone SV. Reduced prevalence of AD in users of NSAIDs and H2 receptor antagonists: the Cache County study. Neurology. 2000 Jun 13;54(11):2066-71. doi: 10.1212/wnl.54.11.2066. PMID 10851364
- [Background] Breitner JC. The role of anti-inflammatory drugs in the prevention and treatment of Alzheimer's disease. Annu Rev Med. 1996;47:401-11. doi: 10.1146/annurev.med.47.1.401. PMID 8712791
- [Background] McGeer PL, Schulzer M, McGeer EG. Arthritis and anti-inflammatory agents as possible protective factors for Alzheimer's disease: a review of 17 epidemiologic studies. Neurology. 1996 Aug;47(2):425-32. doi: 10.1212/wnl.47.2.425. PMID 8757015
- [Result] ADAPT Research Group; Lyketsos CG, Breitner JC, Green RC, Martin BK, Meinert C, Piantadosi S, Sabbagh M. Naproxen and celecoxib do not prevent AD in early results from a randomized controlled trial. Neurology. 2007 May 22;68(21):1800-8. doi: 10.1212/01.wnl.0000260269.93245.d2. Epub 2007 Apr 25. PMID 17460158
- [Result] ADAPT Research Group. Cardiovascular and cerebrovascular events in the randomized, controlled Alzheimer's Disease Anti-Inflammatory Prevention Trial (ADAPT). PLoS Clin Trials. 2006 Nov 17;1(7):e33. doi: 10.1371/journal.pctr.0010033. PMID 17111043
- [Derived] Drye LT, Casper AS, Sternberg AL, Holbrook JT, Jenkins G, Meinert CL. The transitioning from trials to extended follow-up studies. Clin Trials. 2014 Dec;11(6):635-47. doi: 10.1177/1740774514547396. Epub 2014 Aug 12. PMID 25115882
- [Derived] ADAPT-FS Research Group. Follow-up evaluation of cognitive function in the randomized Alzheimer's Disease Anti-inflammatory Prevention Trial and its Follow-up Study. Alzheimers Dement. 2015 Feb;11(2):216-25.e1. doi: 10.1016/j.jalz.2014.03.009. Epub 2014 Jul 9. PMID 25022541
- [Derived] ADAPT Research Group; Martin BK, Szekely C, Brandt J, Piantadosi S, Breitner JC, Craft S, Evans D, Green R, Mullan M. Cognitive function over time in the Alzheimer's Disease Anti-inflammatory Prevention Trial (ADAPT): results of a randomized, controlled trial of naproxen and celecoxib. Arch Neurol. 2008 Jul;65(7):896-905. doi: 10.1001/archneur.2008.65.7.nct70006. Epub 2008 May 12. PMID 18474729
- [Derived] Solomon SD, Wittes J, Finn PV, Fowler R, Viner J, Bertagnolli MM, Arber N, Levin B, Meinert CL, Martin B, Pater JL, Goss PE, Lance P, Obara S, Chew EY, Kim J, Arndt G, Hawk E; Cross Trial Safety Assessment Group. Cardiovascular risk of celecoxib in 6 randomized placebo-controlled trials: the cross trial safety analysis. Circulation. 2008 Apr 22;117(16):2104-13. doi: 10.1161/CIRCULATIONAHA.108.764530. Epub 2008 Mar 31. PMID 18378608